CLINICAL TRIAL: NCT05552287
Title: Prospective Analysis of Pharmacokinetic Infliximab Data in Pediatric CD Patients (ProRAPID)
Brief Title: Pharmacokinetic Infliximab Data in Pediatric Crohn's Disease
Acronym: ProRAPID
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Lissy de Ridder, Medical Doctor; Associate Professor, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProRAPID
Record Dates: First submitted 2022-07-11; First posted 2022-09-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease; Child, Only; Biologic; Inadequate
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intensified induction scheme with Infliximab (Experimental): Intensified induction scheme with Infliximab. IFX will be given intravenously at 10 mg/kg at week 0, and 5 mg/kg at weeks 2, 4, and 8 to all patients (induction). Maintenance will start at week 12, and then ideally continue every 6 weeks.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — IFX will be given intravenously at 10 mg/kg at week 0, and 5 mg/kg at weeks 2, 4, and 8 to all patients (induction). Maintenance will start at week 12, and then ideally continue every 6 weeks till week 24 (end of study). IFX trough levels will be measured at weeks 4, 12, and 24. During the maintenance, the IFX dose and/or interval adjustments, the IFX discontinuation or the start of a co-medication (i.e., an immunomodulator) will be possible on indication (i.e., primary nonresponse, secondary loss of response, intolerance to study medication) at the physicians' discretion.

SUMMARY:
Rationale: Crohn's disease (CD) is a chronic, debilitating inflammatory bowel disease (IBD) which is diagnosed during childhood in up to one in ten patients. The use of anti-tumor necrosis factor (TNF)-α agents has significantly ameliorated CD management. Infliximab (IFX) is the first anti-TNF-α agent registered for pediatric CD. The current dosing recommendation of IFX is extrapolated from adult studies, and it is a weight-based dose (5 mg/kg) delivered during induction (infusion at weeks 0, 2, and 6) and maintenance (every 8 weeks). However, pediatric patients have a 25-40% lower drug exposure compared to adults, particularly children under 10 years of age, resulting in diminished efficacy and an increased risk of developing a complicated disease course. The investigators hypothesize that an intensified IFX induction scheme (instead of the current dosing recommendation) is more effective in the treatment of pediatric CD patients.

Objective: The primary study objective of our study is to assess the efficacy of an IFX intensified induction scheme vs. a standard dosing schedule in improving drug exposure without treatment escalation in pediatric CD patients. Secondary objectives are clinical and biochemical remission without treatment escalation, development of antibodies to IFX (ATI) and adverse reactions.

Study design: An international, multicenter, prospective, open-label trial. Study population: Anti-TNF-α naïve children (age 1-15 years) with CD and an indication to start IFX treatment.

Intervention: IFX will be given intravenously at 10 mg/kg at week 0, and 5 mg/kg at weeks 2, 4, and 8 to all patients (induction). Maintenance will start at week 12, and then ideally continue every 6 weeks till week 24 (end of study). IFX trough levels will be measured at weeks 4, 12, and 24. During the maintenance, the IFX dose and/or interval adjustments, the IFX discontinuation or the start of a co-medication (i.e., an immunomodulator) will be possible on indication (i.e., primary nonresponse, secondary loss of response, intolerance to study medication) at the physicians' discretion. Follow-up will continue for the duration of the study (week 24).

Main endpoint: Proportion of patients with IFX TL ≥ 5 µg/mL at week 12 without treatment escalation.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Definition of the problem

Crohn's disease (CD) is a chronic, debilitating inflammatory bowel disease (IBD) which is diagnosed during childhood in up to one in ten patients. Pediatric CD patients often have more severe and extensive disease compared to adults. Prospective studies in pediatric CD are scarce; therefore, many questions remain unanswered in the treatment of pediatric CD. The discovery of anti-tumor necrosis factor (TNF)-α agents opened up a new window in the pharmacological management of this condition. Infliximab (IFX) was the first anti-TNF-α agent to be approved for use in the treatment of CD. Several clinical studies showed its efficacy in inducing mucosal healing and improving long-term outcomes, even as a first-line treatment. Efficacy of IFX has been related to IFX trough levels, which are dependent on clearance of IFX. Lower IFX trough levels (TLs) are associated with increased immunogenicity and increased risk of developing complicated disease course of time. The clearance of IFX is influenced by many factors. Clearance of IFX in IBD can be influenced by disease severity (i.e., local vs. systemic inflammation), increased intestinal permeability, increased proteatic activity, the presence of antibodies to IFX (ATI), and the use of a concomitant immunomodulatory. Furthermore, the study of Dotan el al. showed that clearance of IFX is not linearly related weight, meaning that patients with lower body weight might need higher IFX doses.

Despite these data, the current dosing recommendation of IFX is still a weight-based dose (5 mg/kg) during induction (infusion at weeks 0, 2, and 6) and the maintenance phase (every 8 weeks) extrapolated from adult studies. However, recent evidence indicates that pediatric patients have a 25-40% lower drug exposure compared to adults. Particularly in children under 10 years of age, Jongsma et al. showed in a retrospective cohort a median IFX TLs at week 14 of 3.1 µg/mL in a subset of young CD patients (age < 10 years), which is far below the recently recommended target trough level > 5 µg/mL at week 14. Based on this data, young children probably need higher IFX dosing to obtain optimal IFX trough levels.

However, up till now no prospective trials have been performed using an intensified dosing scheme for younger CD patients. As stated above, adult data on intensified dosing schemes cannot be directly extrapolated to children due to pharmacokinetic differences. Therefore, a prospective trial within children with CD is necessary to identify a possible new dosing scheme for these patients. This study is innovative, as it will be the first prospective trial to determine if an IFX intensified induction scheme is more effective than standard dose in pediatric CD. This study will provide additional knowledge whether an intensified induction scheme in younger patients will indeed result in higher trough levels and better disease outcomes.

OBJECTIVES

The purpose of this study is to define an optimal IFX dosing schedule for patients aged 1-15 years with CD.

The primary study objective is:

- To assess the proportion of patients with IFX Trough level ≥ 5 µg/mL at week 12 without treatment escalation

The secondary objectives are:

* To assess the efficacy of an IFX intensified induction scheme in obtaining clinical and biochemical remission at weeks 4, 12, and 24 without treatment escalation.
* To assess whether an intensified induction scheme increases the frequency of ATI and/or of infusion reactions/adverse reactions.
* To assess factors that will predict who will respond to IFX based on proteomic analysis.

STUDY DESIGN

The investigators will perform an international, multicenter, prospective, open-label trial. The study duration for each individual participant will consist of a 4-week screening period and a 24-week intervention period. Patients will be enrolled over 12 months. The study will be completed in 24 months. An illustration of the study design is given in supplement 1.

STUDY POPULATION

Approximately 50 patients aged 1-15 years (30 patients aged 1-9 years and 20 patients aged 10-15 years) with CD and an indication to start IFX will be prospectively enrolled. Patients will be recruited in academic centers with specific expertise in pediatric IBD within Europe.

TREATMENT OF SUBJECTS

Investigational treatment

IFX will be given intravenously at 10 mg/kg at week 0, and 5 mg/kg at weeks 2, 4, and 8 to all patients (induction). Maintenance will start at week 12, and then ideally continue every 6 weeks. The choice of this intensified induction scheme was based on both preliminary modeling and experience gained from everyday clinical practice. The investigational medicinal product is infliximab (Inflectra®, Hospira, or any of the other biosimilars of IFX according to the local availability in the participating centre) administered intravenously with a more intensified induction scheme.

Use of co-intervention at the start of IFX

Patients are allowed to enter the study if they receive other drugs (co-medications) at the start of IFX. The allowed co-medications and their restrictions are as follows:

* Steroids: when started more than 2 weeks before the first IFX infusion. Patients will be instructed to follow a tapering schedule aiming at corticosteroid withdrawal by week 12.
* Mesalazine: when started more than 2 weeks before first IFX infusion, the dose should not be increased through week 24.
* EEN: when started more than 2 weeks before the first IFX infusion
* Partial Enteral Nutrition, Crohn's Disease Exclusion Diet or other dietary therapy
* Azathioprine (AZA) or methotrexate (MTX): the dose should not be increased through week 24 except for weight-based or metabolite-based adjustments. AZA/MTX can be discontinued at any time.

Escape medication

During the follow-up, there may be a need for an additional CD-related intervention, which may be indicated in the case of primary non-response, secondary LOR, or intolerance to study medication. In these situations, treatment changes will be made at the physicians' discretion, and follow-up will continue for the duration of the study (week 24).

Allowed additional CD-related treatment may be:

* Increasing dose of IFX (advised) or shortening of the interval
* Start or intensification of Exclusive or polymeric enteral nutrition
* Start or intensification of steroids (oral or topical)
* Start or intensification of immunomodulators (AZA, MTX) (except intensification based on weight or metabolites).
* Start or intensification of mesalazine (oral or topical)
* Start of antibiotics (limited to indication for CD, i.e. perianal disease)
* Start of biologics other than anti-TNF-α (including but not limited to ustekinumab, vedolizumab, abatacept, anakinra, etc.)
* Start of other CD related treatment specified in the European guideline of CD in children.

Study procedures

Screening for eligible participants will be performed within 4 weeks prior to the first IFX infusion. Before starting IFX, as part of usual clinical care patients will be screened for the following infections: tuberculosis, hepatitis B and C and Epstein-Barr virus.

If patients are included within the study, they will undergo the following study procedures:

* IFX will be given intravenously at 10 mg/kg at week 0, and 5 mg/kg at weeks 2, 4, and 8 to all patients (induction). Maintenance will start at week 12, and then ideally continue every 6 weeks. The choice of this intensified induction scheme was based on both preliminary modeling and experience gained from everyday clinical practice.
* Study visits will be scheduled at each IFX infusion at week 0 (baseline), 2, 4, 8, 12, and 24 (end of study). At each visit, the following parameters will be assessed: clinical disease activity (wPCDAI), weight (kg), height (cm), concomitant medication (type and dosage), IFX dosage and interval, changes in medication, adverse events, and IBD standard laboratory tests (hemoglobin, hematocrit, white blood cells, platelet count, CRP, erythrocyte sedimentation rate - ESR, albumin). wPCDAI is a validated instrument for measuring disease activity in children and adolescents with CD. This score is a mathematically weighted version of PCDAI. The wPCDAI is composed of three domains (clinical symptoms, physical examination, and laboratory variables), with individual items mathematically weighted to produce an overall score that classifies patients into 4 disease activity categories: none, < 12.5; mild, 12.5 to 40; moderate, > 40 to 57.5; and severe, > 57.5. A decrease of 17.5 points is taken as evidence of improvement.
* IFX TLs will be measured at weeks 4, 12, and 24. ATI will be measured if IFX TL < 1 µg/mL. Blood samples will be taken to determine IFX TLs and ATI. All blood samples will be taken during a routine blood draw or out of the already inserted infusion needle. For the purpose of this study, one extra tube of blood will be drawn. Blood samples for TLs and ATI will be locally stored at -80 °C and then sent to the coordinating center (Erasmus MC) to be analyzed (ELISA assay). On clinical indication, IFX TLs and ATI can also be determined locally in the participating centers.
* FC (quantitative) will be measured at baseline, week 12 and 24. FC is a non-invasive tool to evaluate mucosal healing. Assays for FC concentration will be performed using a validated method at study site laboratories.
* Quality of life will be checked in order to assess the impact on quality of life of the intensified induction scheme. It will be assessed at baseline, weeks 12, and 24. Quality of life will be assessed with the IBD-specific Impact-III score and EQ-5D-Y questionnaire.

The total duration of follow-up will be 24 weeks. During the follow-up, the IFX dose and/or interval adjustments or the IFX discontinuation will be possible on indication (i.e., primary nonresponse, secondary LOR, intolerance to study medication) at the physicians' discretion. Any adjustments will be notified to the coordinating center.

Withdrawal of individual subjects

No specific criteria for study withdrawal exist. Patients can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons. The treating physician can deviate from the study protocol for medical reasons (i.e., persistent non-response or LOR despite adequate IFX TLs and treatment escalation, high ATI, severe infusion reactions, severe adverse reactions).

STATISTICAL ANALYSIS

Parametric variables will be described by their mean and standard deviation (SD) and compared with use of the T-test. Non-parametric variables will be described by their median and interquartile range and compared using the Mann-Whitney U test. Categorical variables will be summarized using counts and percentages. A Chi-squared test will be used for analyses without a stratification factor. All statistical testing will be 2-sided and significant at the 0.05 level. Missing data will be reported and left out of analyses. Graphical data displays (i.e., box plots) may also be used to summarize the data.

Statistical test primary endpoint:

To test whether the percentage in the study group will be different from the population, the one sample Z-test will be performed. In the RAPID cohort, 68% of patients with CD and age <10 had trough levels <5 ug/ml. Null hypotheses will be that percentage of patients with trough level >5 ug/ml without treatment escalation will be similar to (100%-68%=) 32% (based on outcomes of the RAPID cohort). Alternative hypothesis will be that percentage will be different from 32%. The assumptions that will be tested are the following: p · n ≥ 10 and (1 - p) · n ≥ 10. If these assumptions are not met, the proportion of patients reaching the primary endpoint will be tested by the non-parametric one sample Binomial Test.

ELIGIBILITY:
Inclusion Criteria:

* Anti-TNF-α naïve children (age 1-15 years) with CD and an indication to start IFX treatment will be eligible for inclusion after a diagnosis of CD is made based on the Porto criteria. Indications of starting IFX treatment as per ECCO-ESPGHAN guidelines include non-response after induction with exclusive enteral nutrition or steroids, non-response to immunomodulators, severe growth delay, extensive disease and/or structuring or penetrating disease, with or without perianal disease. Evaluation of the indication to start IFX is performed at the discretion of the attending physician.

Exclusion Criteria:

* Established monogenetic IBD
* Diagnosis with UC or IBD-U, ulcerative colitis like
* Active fistulizing/perianal disease at start of IFX treatment (patients with inactive fistulizing/perianal disease are allowed to participate)
* Severe comorbidity (not related to IBD)
* Immediate need for surgery (i.e., symptomatic stenosis or stricture in the bowel)
* Severe infection such as sepsis or opportunistic infections, positive tuberculin test or a chest radiograph consistent with tuberculosis or malignancy
* Pregnancy, suspected or definitive
* Treatment with anti-TNF or other biological drugs in the past
* Start of corticosteroids or mesalazine less than 2 weeks prior to first IFX infusion
* Start of Exclusive Enteral Nutrition less than 2 week prior to first IFX infusion

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with IFX Trough Levels ≥ 5 µg/mL at week 12 without treatment escalation | 12 weeks
  Treatment escalation is defined as any additional CD-related medication or IBD-related abdominal surgery

SECONDARY OUTCOMES:
Proportion of patients with IFX Trough Levels ≥ 5 µg/mL at week 24 without the need for treatment escalation | 24 weeks
  Treatment escalation is defined as any additional CD-related medication or IBD-related abdominal surgery
Clinical and biochemical remission at weeks 4, 12, and 24 without the need for treatment escalation in patients with TL ≥ 5 µg/mL and in patients with TL < 5 µg/mL. | 24 weeks
  Clinical remission is defined as wPCDAI <12.5 Biochemical remission is defined as CRP <5 mg/dL, FC <250 ug/g.
Predictors of IFX Trough Levels at weeks 4, 12, and 24. Factors included in this analysis will be sex, age, body mass index (BMI), wPCDAI, IBD laboratory values, antibodies to Infliximab (ATI), dose, and interval of IFX infusions. | 24 weeks
Development of antibodies to IFX until week 24 | 24 weeks
  ATI's will be assessed if IFX TL is <1 ug/ml at week 4, 12 or 24.
Prediction of reponders versus non-responders to IFX based on proteomic analysis. | 24 weeks
  Responders will be defined as decrease of 17.5 in wPCDAI at week 6 from start of IFX. Serum immune proteins will be analysed using the OLINK technique. It will be investigated whether there are predictive immune proteins of IFX response
Evaluation of quality of life | 24 weeks
  Quality of life will be assessed at baseline, weeks 12 and 24 in all patients.

OTHER OUTCOMES:
Proportions of patients with primary non-response | 24 weeks
  Primary non-response: absence of response (wPCDAI decrease > 17.5) at week 6 compared to baseline
Proportions of patients with secondary loss of response (LOR) | 24 weeks
  Secondary LOR: either an increase in wPCDAI > 17.5 or a total wPCDAI score > 40 in a patient who previously responded to induction treatment rates over time.
Evaluation of number of adverse events | 24 weeks
  Adverse event rate over time.Adverse events are defined as any undesirable experience occurring to a subject during the study, whether considered related to the investigational product or not. All adverse events reported spontaneously by the subject or observed by the investigator, or his staff will be recorded.
Complications rate | 24 weeks
  Complication rate (fistulas, abscesses, strictures, surgery, extraintestinal manifestations) over time.
Baseline demographics | 24 weeks
  Age at diagnosis, age at start of IFX, ethnicity, sex, weight, height
Baseline clinical covariates | 24 weeks
  Reason for starting IFX, Paris classification, concomitant drugs, IBD standard laboratory values (haemoglobin, haematocrit, leukocytes, thrombocytes, CRP, ESR, albumin), faecal calprotectin, wPCDAI score, comorbidity/extra-intestinal manifestations and, if available, magnetic resonance imaging and the simple endoscopic score for CD (SES-CD).
Cost-effectiveness analysis of costs of treatment versus quality of life. | 24 weeks
  In consultation with Department of Economics and Health, calculation of costs per QALY based on quality of life questionnaires will be made.
Height | 24 weeks
  Height will be measured in centimeters
Weight | 24 weeks
  Weight will be measured in kilograms
Body Mass Index | 24 weeks
  Height and height will be combined to report BMI in kg/m^2
IMPACT-III | 24 weeks
  Disease-specific quality of life will be obtained with the IMPACT-III questionnaire (range 0-100) in patients (≥9 years old) at week 0, 12 and 24. A higher score indicates a higher quality of life. The questionnaire consists of 35 items encompassing 6 domains: bowel symptoms, systemic symptoms, emotional functioning, social functioning, body image and treatment/interventions
EQ-5D-Y | 24 weeks
  Quality of life will be obtained with the EQ-5D-Y questionnaire. This questionnaire consists of 5 dimensions (range 1-3 per dimension) and a Visual Analogue Scale (range 0-100).
Age | 24 weeks
  In years
Weighted Paediatric Crohn's disease activity index (wPCDAI) | 24 weeks
  This is a clinical disease activity score with range 0-125. A higher score indicates worse disease activitiy.
Dose of Infliximab in miligrams | 24 weeks
Haemoglobin in mmol/L | 24 weeks
Haematocrit in L/L | 24 weeks
CRP in mg/L | 24 weeks
ESR in mm/h | 24 weeks
Thrombocytes x 10^9/L | 24 weeks
Leukocytes x 10^9/L | 24 weeks
Albumin in g/L | 24 weeks
Faecal calprotectin in ug/g | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lissy de Ridder, PhD, Principal Investigator — Erasmus Medical Center - Sophia Children's Hospital
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No